CLINICAL TRIAL: NCT01787565
Title: Pilot Evaluation to Assess the Clinical and Economic Impact of Pfizer's Pain Management Program (painPREMIER) in the Treatment of Low Back Pain, in an Occupational Health Care Setting in Finland
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Collaborators: Terveystalo (Other)
Responsible Party: Sponsor
Other Study IDs: X9001016
Record Dates: First submitted 2013-01-22; First posted 2013-02-08 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Back Pain
Keywords: non-interventional; clinical; investigation; low; back; pain; painPREMIER
MeSH Terms: conditions — Back Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- painPREMIER cohort
  Interventions: Other: painPREMIER cohort
- Control cohort
  Interventions: Other: Control cohort

INTERVENTIONS:
Other: painPREMIER cohort — Low back pain patients prospectively recruited during the study period and managed with painPREMIER.
  Groups: painPREMIER cohort
Other: Control cohort — A matched group of low back pain patients not managed with painPREMIER.
  Groups: Control cohort

SUMMARY:
The aim of this investigation is to determine whether the use of painPREMIER will significantly improve function in patients with low back pain in an occupational health clinical setting. painPREMIER is a tool that assists clinicians in the accurate diagnosis of back pain and associated problems in order to treat them most effectively.

DETAILED DESCRIPTION:
Patients presenting at feeder sites to be referred to low back pain clinic and assessed for eligibility A decision was made to terminate this study on 09 OCT 2013. The study was terminated for operational/business reasons. This study was not terminated for reasons of safety or efficacy.

ELIGIBILITY:
Inclusion Criteria:

* New episode of low back pain
* Member of Terveystalo health insurance scheme

Exclusion Criteria:

* Previous back pain related healthcare visit in the last 3 months
* Patients identified as having a 'red flag' condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Members of the Terveystalo health insurance scheme presenting with a new episode of low back pain
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire | 3 months
  Change from baseline

SECONDARY OUTCOMES:
Roland Morris Disability Questionnaire | 6 months
  Change from baseline
Self-reported low back pain intensity | 3 months
  Change from baseline
Self-reported low back pain intensity and Roland Morris Disability Questionnaire | 3 months
  Proportion of patients with at least 30% and 50% improvement
Global Assessment of Disease Activity | any time up to 6 months
  Change from baseline
SF-12 (Short Form 12 Health Survey), v2.0 (Mental Component Summary Scale and Physical Component Summary Scale) | 3 months
  Change from baseline
EQ5-D Health Questionnaire | 3 months
  Change from baseline
PHQ-4 (Patient Health Questionnaire for Depression and Anxiety-4) | 3 months
  Proportion of patients at risk for depression and/or anxiety
Self-reported depression PHQ-8 (Patient Health Questionnaire for Depression and Anxiety-8) and anxiety GAD-7 (Generalized Anxiety Disorder 7-item scale) | 3 months
  Changes from baseline (if collected at BL)
Self-reported catastrophizing - Coping Strategies Questionnaire - Catastrophizing scale (CSQ-CAT) | 3 months
  Changes from baseline
Self-reported absenteeism, presenteeism, lost productivity and activity, over prior 2 weeks, measured by Work Productivity and Activity Impairment (WPAI): Specific Helath Problem (Low Back Pain) questionnaire (painPREMIER cohort) | 3 months
  Changes from baseline
All-cause absence days and costs associated with sick leave | 3 months
  Comparison between painPREMIER cohort and control cohort
All-cause pharmacy and medical resource use/costs | 3 months
  Comparison of pre and post-enrollment for both cohorts
Low back pain-related medical resource use/costs and pharmacy use/costs | 3 months
  Comparison of pre and post-enrollment for both cohorts
Low back pain-specific medical resource use/costs | 3 months
  Comparison of pre and post-enrollment for both cohorts
Total low back pain direct medical costs | 3 months
  Comparison of pre and post-enrollment for both cohorts
Overall low back pain costs via claims data and imputed WPAI:LBP Work Productivity and Activity Impairment (WPAI): Specific Helath Problem (Low Back Pain) questionnaire | 3 months
  Comparison between painPREMIER and control cohort
Overall all costs via claims and absence data | 3 months
  Comparison between painPREMIER and control cohort
Patient Satisfaction | 3 months
  Patient Satisfaction with painPREMIER
Specialist Occupational Health Provider Satisfaction | After enrolment complete estimated 4 months
  Specialist Occupational Health Provider Satisfaction with painPREMIER
Net Promoter Score | 1 week
  Net Promoter Score
Semi-structured interview | 6 months
  Patient feedback
Specialist Occupational Health Provider Engagement | 6 months
  Specialist Occupational Health Provider Engagement with portal
Specialist Occupational Health Provider treatment recommendations | 6 months
  Specialist Occupational Health Provider treatment recommendations vs painPREMIER treatment recommendations
Patient engagement/treatment adherence | 6 months
  Platform use, CBST(Cognitive Behavioral Skills Training) module use and adherence to pharmacological therapy
TAMPA17 Scale for Kinesiophobia, PHQ4, PHQ8, (Patient Health Questionnaire for Depression and Anxiety-4 and 8), GAD7 (Generalized Anxiety Disorder 7-item scale) | Baseline
  To evaluate the correlation between TAMPA17, PHQ4, PHQ8, GAD7 baseline assessments in the painPREMIER cohort
painDETECT, TAMPA17 Scale for Kinesiophobia, LBPI (low back pain intensity) and RMDQ (Roland Morris Disability Questionnaire) | 3 months
  To evaluate the change from baseline and correlation between the instruments in the painPREMIER cohort
Sub-group analysis | 6 months
  To evaluate patterns of use and outcomes in subgroups
Daily sleep intereference rating scale | 3 months
  Change from baseline
Daily sleep intereference rating scale | 6 months
  Change from baseline
Self-reported low back pain intensity and Roland Morris Disability Questionnaire | 6 months
  Proportion of patients with at least 30% and 50% improvement
SF-12 (Short Form 12 Health Survey), v2.0 (Mental Component Summary Scale and Physical Component Summary Scale) | 6 months
  Change from baseline
EQ5-D Health Questionnaire | 6 months
  Change from baseline
PHQ-4 (Patient Health Questionnaire for Depression and Anxiety-4) | 6 months
  Proportion of patients at risk for depression and/or anxiety
Self-reported depression PHQ-8 (Patient Health Questionnaire for Depression and Anxiety-8) and anxiety GAD-7 (Generalized Anxiety Disorder 7-item scale) | 6 months
  Changes from baseline (if collected at BL)
Self-reported catastrophizing (CSQ-CAT) Coping Strategies Questionnaire - Catastrophizing scale | 6 months
  Change from baseline
Self-reported absenteeism, presenteeism, lost productivity and activity, over prior 2 weeks, measured by Work Productivity and Activity Impairment (WPAI): Specific Helath Problem (Low Back Pain) questionnaire (painPREMIER cohort) | 6 months
  Changes from baseline
All-cause absence days and costs associated with sick leave | 6 months
  Comparison between painPREMIER cohort and control cohort
All-cause pharmacy and medical resource use/costs | 6 months
  Comparison of pre and post-enrollment for both cohorts
Low back pain-related medical resource use/costs and pharmacy use/costs | 6 months
  Comparison of pre and post-enrollment for both cohorts
Low back pain-specific medical resource use/costs | 6 months
  Comparison of pre and post-enrollment for both cohorts
Total low back pain direct medical costs | 6 months
  Comparison of pre and post-enrollment for both cohorts
Overall low back pain costs via claims data and imputed WPAI:LBP Work Productivity and Activity Impairment (WPAI): Specific Helath Problem (Low Back Pain) questionnaire | 6 months
  Comparison between painPREMIER and control cohort
Overall all costs via claims and absence data | 6 months
  Comparison between painPREMIER and control cohort
Patient Satisfaction | 6 months
  Patient Satisfaction with painPREMIER
Net Promoter Score | 3 months
  Net Promoter Score

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Helsinki, Finland

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=X9001016